CLINICAL TRIAL: NCT03480087
Title: Subclinical Cardio-toxicities Evaluation With Strain Rate Echocardiography After Chemotherapy and/or Mediastinal Radiotherapy in Patient With Lymphoma
Acronym: Cardiocare
Status: Completed | Type: Observational
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Mario Levis, Medical doctor, A.O.U. Città della Salute e della Scienza
Other Study IDs: Cardiocare
Record Dates: First submitted 2018-03-14; First posted 2018-03-29 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Lymphoma, Non-Hodgkin; Hodgkin Lymphoma; Toxicity, Cardiac
Keywords: strain-rate echocardiography; chemotherapy; radiotherapy, mediastinal; Lymphoma; Hodgkin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease; Cardiotoxicity; Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chemotherapy alone: Patient treated with anthracycline containing chemotherapy
- Chemotherapy plus radiotherapy: Patient treated with anthracycline containing chemotherapy followed by mediastinal radiotherapy

SUMMARY:
Treatments-related cardiotoxicity is a critical issue in long term lymphoma survivors, particularly at young age, and its early identification is important to prevent clinically relevant cardiac events. Complete echocardiographic assessment including 2-dimension global longitudinal strain (2D-GLS), seems to be an effective tools in detecting preclinical systolic changes to the cardiac function even when the ejection fraction is preserved. The aim of Cardiocare study is to investigate early detection of subclinical chemo and radiation-induced changes in left ventricular function using 2D-GLS.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Diagnosis of Hodgkin Disease (HD) or Primary Mediastinal B-cell lymphoma (PMBCL) or diffuse large B-cell lymphoma (DLBCL)
* Disease requiring treatment with anthracycline containing regimen only (cohort A) or anthracycline containing regimen followed by mediastinal radiotherapy (cohort B)
* Written informed consent

Exclusion Criteria:

* Age > 70 years
* Unable to perform anthracyline containing regimen
* Previous treatment with mediastinal radiotherapy
* Kidney failure (defined as creatinine x2 UNL) or liver failure (defined as AST and ALT x2 UNL)
* ECOG PS > 2
* Echocardiographic acoustic windows not suitable for strain evaluation
* Any other conditions or situations preventing patients to sign informed consent

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient 19-70 years old with HD or PMBCL or DLBCL requiring treatment with chemotherapy or chemotherapy plus mediastinal radiotherapy suitable for a strain-rate echocardiograpy evaluation
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2022-07 (Actual); Study Completion 2022-07 (Actual)

PRIMARY OUTCOMES:
Left ventricular ejection fraction (LVEF) | Baseline, Change of LVEF from Baseline at 4/6 month (end of chemotherapy), Change of LVEF from Baseline at 6/8 months (end of radiotherapy - if applicable), Change of LVEF from Baseline at 9/11 months (3 months after treatment completion)
  Left ventricular ejection fraction measured by echocardiography
Global Longitudinal Strain (GLS) | Baseline, Change of GLS from Baseline at 4/6 month (end of chemotherapy), Change of GLS from Baseline at 6/8 months (end of radiotherapy - if applicable), Change of GLS from Baseline at 9/11 months (3 months after treatment completion)
  Global Longitudinal Strain measured by strain-rate echocardiography

SECONDARY OUTCOMES:
Anthracycline cumulative dose | 4/6 month after baseline (end of chemotherapy)
  Anthracycline cumulative dose
T troponin | Baseline, Before each chemotherapy administration, 4/6 month after baseline (end of chemotherapy), 6/8 months after baseline (end of radiotherapy - if applicable), 9/11 months after baseline (3 months after treatment completion)
  T troponin rate

CONTACTS AND LOCATIONS:
Locations (1):
- SC Ematologia - AOU Città della salute e della Scienza di Torino, Torino, Italy